CLINICAL TRIAL: NCT04262466
Title: Phase 1/2 Study of IMC-F106C in Advance PRAME-Positive Cancers
Brief Title: Safety and Efficacy of IMC-F106C as a Single Agent and in Combination With Checkpoint Inhibitors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMC-F106C-101
Record Dates: First submitted 2020-01-30; First posted 2020-02-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Select Advanced Solid Tumors
MeSH Terms: interventions — pembrolizumab; Drug Therapy; Antibodies, Monoclonal; tebentafusp; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Brenetafusp Monotherapy (Experimental): Participants receive brenetafusp.
  Interventions: Drug: Brenetafusp
- Brenetafusp and Anti-PD(L)1 Agent (Experimental): Participants receive brenetafusp and pembrolizumab.
  Interventions: Drug: Brenetafusp and pembrolizumab
- Brenetafusp and Chemotherapy (Experimental): Participants receive brenetafusp and chemotherapy. Choice of chemotherapy is dependent on cohort.
  Interventions: Drug: Brenetafusp and chemotherapy
- Brenetafusp and Targeted Therapy (Experimental): Participants receive brenetafusp and a selected targeted therapy. Receipt of kinase inhibitor is dependent on histology.
  Interventions: Drug: Brenetafusp and tebentafusp; Drug: Brenetafusp and bevacizumab; Drug: Brenetafusp and kinase inhibitors
- Brenetafusp and Multimodal Therapy (Experimental): Participants receive brenetafusp, biologics (eg, pembrolizumab, bevacizumab) IV infusions and chemotherapy IV infusions based on histology.
  Interventions: Drug: Brenetafusp and monoclonal antibodies and chemotherapy

INTERVENTIONS:
Drug: Brenetafusp — Brenetafusp IV infusions
  Arms: Brenetafusp Monotherapy
Drug: Brenetafusp and pembrolizumab — Brenetafusp and pembrolizumab IV infusions
  Arms: Brenetafusp and Anti-PD(L)1 Agent
Drug: Brenetafusp and chemotherapy — Brenetafusp and chemotherapy IV infusions
  Arms: Brenetafusp and Chemotherapy
Drug: Brenetafusp and monoclonal antibodies and chemotherapy — Brenetafusp and a monoclonal antibody therapy and chemotherapy
  Arms: Brenetafusp and Multimodal Therapy
Drug: Brenetafusp and tebentafusp — Brenetafusp and tebentafusp IV infusions
  Arms: Brenetafusp and Targeted Therapy
Drug: Brenetafusp and bevacizumab — Brenetafusp and bevacizumab IV infusions
  Arms: Brenetafusp and Targeted Therapy
Drug: Brenetafusp and kinase inhibitors — Brenetafusp and oral kinase inhibitors
  Arms: Brenetafusp and Targeted Therapy

SUMMARY:
Brenetafusp (IMC-F106C) is an immune-mobilizing monoclonal T cell receptor against cancer (ImmTAC ®) designed for the treatment of cancers positive for the tumor-associated antigen PRAME. This is a first-in-human trial designed to evaluate the safety and efficacy of brenetafusp in adult participants who have the appropriate HLA-A2 tissue marker and whose cancer is positive for PRAME.

DETAILED DESCRIPTION:
The IMC-F106C-101 Phase 1/2 study will be evaluated in patients with metastatic/unresectable tumors which include select Advanced Solid Tumors and will be conducted in two phases.

1. Phase 1: To identify the Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 dose (RP2D) of brenetafusp as a single agent and administered in combination with chemotherapies, targeted therapies, and monoclonal antibodies.
2. Phase 2: To assess the efficacy of brenetafusp in selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG PS 0 or 1
2. HLA-A*02:01 positive
3. PRAME positive tumor
4. Relapsed from, refractory to, or intolerant of standard therapies; or, in combination with standard therapies
5. If applicable, must agree to use highly effective contraception

Exclusion Criteria:

1. Symptomatic or untreated central nervous system metastasis
2. Recent bowel obstruction
3. Ongoing ascites or effusion requiring recent drainages
4. Significant immune-mediated adverse event with prior immunotherapy (Participants in checkpoint inhibitor combination treatment)
5. Inadequate washout from prior anticancer therapy
6. Significant ongoing toxicity from prior anticancer treatment
7. Out-of-range laboratory values
8. Clinically significant lung, heart, or autoimmune disease
9. Ongoing requirement for immunosuppressive treatment
10. Prior solid organ or bone marrow transplant
11. Active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection
12. Significant secondary malignancy
13. Hypersensitivity to study drug or excipients
14. Antibiotics, vaccines or surgery within 2-4 weeks prior to the first dose of study intervention
15. Pregnant or lactating participants
16. Any other contraindication for applicable combination partner based on local prescribing information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 727 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of dose-limiting toxicity (DLT)s | Up to ~28 days after each dose
Phase 1: Incidence of adverse events (AE) and serious adverse events (SAE) | Up to 30 days after the last dose of study therapy
Phase 1: Number of participants with dose interruptions, dose reductions, or dose discontinuations | Up to ~12 months
Phase 1: Number of participants with abnormal laboratory test results (hematology) | Up to 30 days after the last dose of study therapy
Phase 1: Number of participants with abnormal laboratory test results (chemistry) | Up to 30 days after the last dose of study therapy
Phase 1: Number of participants with abnormal laboratory test results (coagulation) | Up to 30 days after the last dose of study therapy
Phase 1: Number of participants with abnormal urinalysis | Up to 30 days after the last dose of study therapy
Phase 1: Number of participants with abnormal vital signs | Up to 30 days after the last dose of study therapy
Phase 1: Mean change from baseline in QTcF interval | Up to 30 days after the last dose of study therapy
Phase 2: Best overall response (BOR) | Up to ~2 years

SECONDARY OUTCOMES:
Phase I: Best Overall Response (BOR) | Up to ~2 years
Progression-free survival (PFS) | Up to ~2 years
Duration of response (DOR) | Up to ~2 years
Overall survival | Up to ~2 years
Area under the plasma concentration-time curve (AUC) of brenetafusp | At designated time points up to ~3 weeks
Maximum plasma drug concentration (Cmax) of brenetafusp | At designated time points up to ~3 weeks
Time to reach maximum plasma concentration (Tmax) of brenetafusp | At designated time points up to ~3 weeks
Plasma elimination half-life (t½) of brenetafusp | At designated time points up to ~3 weeks
Incidence of anti-brenetafusp antibody formation | Up to ~ 2 years
Changes in lymphocyte counts over time | Up to ~3 weeks
Changes in serum cytokines over time | Up to ~3 weeks
Local tumor response based on Gynecological Cancer Intergroup (GCIG) Cancer Antigen 25 (CA-125) response criteria | Up to ~2 years

CONTACTS AND LOCATIONS:
Locations (76):
- United States (22):
  - University of California - San Diego, La Jolla, California
  - Angeles Clinic and Research Institute, Los Angeles, California
  - University of California Davis Comprehensive Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Houston Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (4):
  - Scientia Clinical Research, Randwick, New South Wales
  - Melanoma Institute Australia (MIA) - The Poche Centre, Wollstonecraft, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- LKH - Universitätsklinikum der PMU Salzburg, Salzburg, Austria
- Belgium (6):
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - CHU de Liege, Liège, Luik
  - Institut Jules Bordet, Brussels
  - UZA, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (4):
  - Hospital Nossa Senhora da Conceicao, Porto Alegre
  - D'Or Institute for Research and Education, Rio de Janeiro
  - National Cancer Institute, Rio de Janeiro
  - Hospital Israelita Albert Einstein, São Paulo
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM Centre de Recherche, Montreal, Quebec
- France (5):
  - Institut Bergonie - Nouvelle-Aquitaine, Bordeaux, Gironde
  - Gustave Roussy (Institut de Cancerologie Gustave-Roussy), Villejuif, Val De Marne
  - Universite Claude Bernard Lyon Est, Lyon, Villeurbanne
  - Hopital Saint-Louis - Centre d'Onco-Dermatologie, Paris
  - Institut Curie, Paris
- Universitaetsklinikum Heidelberg, Heidelberg, Germany
- St Vincents University Hospital, Dublin, Ireland
- Italy (3):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Dipartimento di Medicina Interna e Scienze Mediche, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Patologia Ostetrica e Ginecologica, Seriate, Roma
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale, Napoli
- Netherlands (3):
  - Netherlands Cancer Institute, Amsterdam, CX
  - UMC Groningen Comprehensive Cancer Center, Groningen, GZ
  - Leiden UMC, Leiden, ZA
- New Zealand Clinical Research-Auckland, Auckland, New Zealand
- Poland (2):
  - Centrum Medyczne Pratia Poznan - Skorzewo, Skórzewo
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Yonsei University College of Medicine, Seoul
  - University of Ulsan College of Medicine, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Universidad de Navarra - Clinica Universidad de Navarra (CUN) - Pamplona, Pamplona, Navarre
  - NEXT Barcelona, Barcelona
  - Hospital Universitario Vall dHebron, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Universidad de Navarra - Clinica Universidad de Navarra (CUN) - Madrid, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
- Switzerland (3):
  - University Hospital, Basel Switzerland, Basel
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne
  - University Hospital of Zurich, Zurich
- United Kingdom (8):
  - Sarah Cannon Research Institute UK, London, City of London
  - University of Oxford, Oxford, Oxfordshire
  - The Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - University of Liverpool, Liverpool
  - University College Hospital London, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital, Surrey Quays